CLINICAL TRIAL: NCT07010991
Title: Effectiveness of Artificial Intelligence Based Educational Approach in Developing Clinical Reasoning Skills in Physiotherapy Students
Brief Title: Effectiveness of Artificial Intelligence Based Educational Approach in Developing Clinical Reasoning Skills
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Simay Akdemir, MSc. Lecturer Physical Therapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MedipolU-SBF-FTR-SA-01
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-05

CONDITIONS: Student; Student Engagement; Student Education
Keywords: Student; Education; Artificial intelligence; Decision Making

STUDY DESIGN:
Intervention Model Description: A prospective, randomized, controlled educational intervention study to be conducted with the participation of undergraduate students. Participants will be divided into two groups as ChatGPT supported problem-based learning and traditional learning group and will be included in a total of 4 hours of training process on chronic low back pain and rehabilitation, 2 hours per week for 2 weeks. 40 students will be included in the study based on voluntary participation. Basic demographic, academic and technological competence information will be collected from the students who will participate in the study. Collected data will be used to assess equality in comparisons between groups, to define sample characteristics, and to support subgroup analyses when necessary. Students will be divided into small groups of 4-5 people after the initial LBP course and will be asked to study for week and actively participate in the discussion presentations and practice session the following week.
Who Masked: Participant, Investigator
Masking Description: Different educators will be giving the educative courses to the groups without knowing the participants of the other group. And one independent observer will observe the student's decision making processes during the courses.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ChatGPT supported problem-based learning (Active Comparator): Students will be divided into small groups of 4-5 after the initial educative course of low back pain (LBP) by a different instructor. Afterwards, each group will work on chronic LBP case scenarios combined with ChatGPT. Students will engage in discussions on interactive learning, physical development planning, exercise recommendations, and biopsychosocial treatment development with ChatGPT.
  Data obtained from ChatGPT will be reviewed by the instructor for academic accuracy. Students will be actively involved in the discussion presentation and practice session. During the course, question sets created by students and answers obtained from ChatGPT are discussed within the group, prepared for class presentation and feedback is given by the instructor in terms of accuracy, timeliness and scientific relevance.
  Interventions: Other: AI based clinical problem solving education
- Traditional learning group (Active Comparator): Students will watch classical case presentations structured by the instructor and will passively/actively participate in discussions conducted on the case. Information transfer will be instructor-centered, ChatGPT or similar AI-supported tools will not be used in this group. Physical assessment and exercise practices will be carried out with the instructor's direct demonstration and students will take turns in the roles of practitioners or observers. Both groups will be provided with basic resource book chapters, videos and supporting materials on a weekly basis. The lessons will be conducted by an experienced physiotherapist academic and the groups will work with different instructor. Physical assessment and exercise practices will be carried out with the direct demonstration of the instructor, and students will take turns in the roles of practitioners and observers.
  Interventions: Other: Traditional Low Back Pain Education

INTERVENTIONS:
Other: AI based clinical problem solving education — This direct involvement of AI and educators aims to improve learning outcomes by leveraging the scalability of AI and the expertise of educators. The question sets created by students and the answers obtained from ChatGPT are discussed within the group and prepared for class presentation, and the instructor provides feedback on accuracy, timeliness, and scientific relevance. This process aims to support students' participation as active questioners and analyzers, rather than passive consumers of information. Intervention will last for 2 weeks, 2 hours of courses each week, in total 4 hours of education will be given. First 2 hours will be the usage parameters and the knowledge about the ChatGPT system and the 2nd week's 2 hours of education will include the presentations and interactive discussion about the case.
  Arms: ChatGPT supported problem-based learning
Other: Traditional Low Back Pain Education — The first session will be given by an independent/different instructor about the definition, reasons, evaluation and the treatment of low back pain for 2 hours. Afterwards the students will be informed about the content of the next week's interactive course and supplied with the study sources like book, articles by the other lecturer. A week will be given to the students to study and the other week they will meet with the lecturer to discuss over a specific case. At the beginning and end of the courses, outcome measures will taken from the both groups.
  Arms: Traditional learning group

SUMMARY:
In the context of this study, the 2nd and 3rd grade undergraduate students in Medipol University, Department of Physiotherapy and Rehabilitation, will taken into an education program to increase and assess their theoretical knowledge level, clinical decision-making skills and attitudes towards interactive learning with artificial intelligence by applying the ChatGPT-supported PBL module and the results will be compared with traditional teaching methods.

DETAILED DESCRIPTION:
In recent years, the use of artificial intelligence-based applications in the field of health education has been rapidly increasing; especially large language models such as ChatGPT have attracted attention in terms of providing rapid access to information and individualized learning opportunities. Utilizing this potential of artificial intelligence, especially in active learning methods such as problem-based learning (PBL), is seen as an approach that can strengthen student-centered education. It is reported in the literature that ChatGPT-supported learning applications yield positive results in medical education, increase theoretical success and provide significant improvements in clinical skills. However, applications specific to physiotherapy education are still limited in this regard. Physiotherapy education requires students to have not only theoretical knowledge but also versatile skills such as clinical decision-making, problem-solving, and patient communication. Therefore, it is important to systematically investigate the effect of ChatGPT-supported PBL applications on student performance and satisfaction. Professionals should be able to benefit from these systems when they do not know where to start in a different case, and students should be informed about this issue by academicians who are experts in their fields in the university environment. In order to prevent the misuse of these systems, it is thought that academicians should not avoid technology and should benefit from the interactive course processing and correct communication opportunities that these systems can create with patients. Today, teaching students how to use technology instead of telling them not to use it is very important for academic success. In this context, the aim of this study is to evaluate the student's theoretical knowledge level, clinical decision-making skills and attitudes towards interactive learning with artificial intelligence and compare them with traditional teaching methods by applying the ChatGPT-supported PBL module to volunteer groups consisting of undergraduate students of Istanbul Medipol University, Department of Physiotherapy and Rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Being an undergraduate student
* Being voluntary to attend to the courses

Exclusion Criteria:

* Not attending to the sessions on time
* Being a 4th grade student who already took and learned the process of clinical problem solving
* Want to recruit to study during the study process

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-09-10 (Estimated)

PRIMARY OUTCOMES:
Theoretical knowledge test | 4 weeks
  A 20-question multiple choice exam will be administered at the beginning of the study after the initial theoretical LBP course and at the end of the 2nd week of training, in total 3 times. With this way, distinguishing the effect of the lecturer's initial education and student's own studies and research will be possible at the analysis. The exams will be compared between groups to assess the intervention effect. The maximum score for the exam will be 100, and a score below 80 will be considered a failing grade.
Mini Clinical Evaluation Exam (Mini-CEX) | 4 weeks
  Participant's history taking, physical assessment and clinical reasoning skills will be observed by an independent assessor using the 9-point Mini-CEX form. Mini-CEX has been widely accepted as an effective and reliable method for assessing clinical skills. It includes student's ability to obtain a patient's history from the patient and family and to perform physical examinations under the guidance of an instructor. The Mini-CEX scoring system uses a nine-point scale and includes seven standards: medical interview skills, physical examination skills, humanistic qualities/professionalism, clinical judgment, counseling skills, organizational efficiency and general clinical competence. The scale ranges from inadequate (1-3 points), satisfactory (4-6 points) to superior (7-9 points). To maintain consistency, all Mini-CEX assessments will be made by a single assessor. The scale is valid and reliable in Turkish.

SECONDARY OUTCOMES:
Student Satisfaction and Attitude Survey | 4 weeks
  Each student will be asked to complete a self-assessment form, where they evaluate their contributions to the group dynamics and their individual learning process, and a peer-assessment form, where they rate the participation levels of their group mates. Students' satisfaction and the impact of using PBL-ChatGPT on their learning experiences will be assessed with a survey developed from a previous study.
Young Internet Addiction Test | 4 weeks
  This scale, which is used to determine the internet usage habits of the participants, was developed by Young in 1998. There is also a Turkish version of the short form consisting of 12 items for quick assessment. The psychometric properties of the questionnaire were studied by Kutlu et al. and it is valid and reliable in Turkish. Participants are scored between 12-60, with score 1 indicating never and score 5 indicating always. High scores indicate a high risk of internet addiction.
Adult Reading Motivation Scale | 4 weeks
  The scale, developed by Schutte and Malouff (2007) to determine adults' reading motivation, consists of 19 items. The scale assesses individuals' reading motivation by asking questions on subheadings such as self, recognition of competence, and reading to be successful in other areas. A score of 1 indicates strongly disagree, a score of 5 indicates strongly agree, and participants receive scores between 19 and 95. High scores indicate high reading motivation and habit. The psychometric properties of the survey were conducted by Yıldız et al. and it is valid and reliable in Turkish.
Artificial Intelligence Self-Efficacy Scale | 4 weeks
  The Artificial Intelligence Self-Efficacy Scale (AISES) will be used to measure participants' perceptions of competence in using artificial intelligence technologies. The scale was developed by Wang and Chuang (2023) and adapted to Turkish by Uyan and Gültekin (2024) to test its validity and reliability. In the Turkish adaptation study, it was confirmed that the scale consisted of four sub-dimensions (assistance, anthropomorphic interaction, comfort and technological competencies) and contained a total of 21 items. The goodness of fit values were found to be at an acceptable level (CFI=0.887, RMSEA=0.084) and Cronbach's alpha values ranged between 0.708 and 0.782 for the sub-dimensions. The scale to be applied to the participants was structured as a 5-point Likert type (1 = Strongly Disagree, 5 = Strongly Agree).

CONTACTS AND LOCATIONS:
Overall Officials: Gülay ARAS BAYRAM, Associate Professor, Study Director — Medipol University İstanbul
Locations (1):
- Medipol University İstanbul, Istanbul, Kavacık Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
This will our own study design conducted by the lecturers in our department. Therefor the IPD will not be shared with the other researchers.

REFERENCES:
- [Derived] Ergezen Sahin G, Aras Bayram G, Sanchez Sierra A, Akdemir S, Kurc D, Tarakci D, Tunali AN. Effects of artificial intelligence based physiotherapy educational approach in developing clinical reasoning skills: a randomized controlled trial. BMC Med Educ. 2025 Oct 9;25(1):1378. doi: 10.1186/s12909-025-07926-w. PMID 41068907